CLINICAL TRIAL: NCT04112537
Title: Dermatologic Clinical Patterns Study of Tuberous Sclerosis Complex Patients Related With Their Somatic Mutation
Brief Title: Dermatologic Patterns of Tuberous Sclerosis Patients and Somatic Mutation Relationship
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0460
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Tuberous Sclerosis Complex
Keywords: Tuberous Sclerosis Complex; MTOR associated protein; Neurocutaneous Syndromes; High-Throughput Nucleotide Sequencing
MeSH Terms: conditions — Tuberous Sclerosis; Neurocutaneous Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Tuberous Sclerosis is a rare genetic disorder that affects about one in 15,000 individuals. It is part of the phacomatoses: a germline mutation of the gene Tuberous Sclerosis Complex 1 (TSC1) or TSC2 causes a protein dysfunction, hamartin and tuberin respectively, leading to mTOR signaling pathway activation, thus tumors rise on the skin but also brain, eyes, kidneys, heart.

Thanks to the advent of sequencing techniques of the human genome, genes involved were found twenty years ago. Most commonly, these are de novo private mutations and autosomal dominant Mendelian transmission. About 15% of patients have a phenotype corresponding to the disease but no mutation is found.

Although the initial clinical description was in 1880, publications regularly describe new signs in Tuberous Sclerosis, especially for skin.

Cutaneous manifestations are important in the diagnostic criteria of the disease and often even the first sign of appeal. However, no data is available on the relationship between genotype and dermatological phenotype.

Therefore the investigator intend to review all cutaneous finding in Tuberous Sclerosis patient and try to link with their mutation.

ELIGIBILITY:
Inclusion criteria:

- Diagnosis of Tuberous Sclerosis Complex established of confirmed by a geneticin, with a genetic study done or processing, patients accepting to be exanimated

Exclusion criteria:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients followed in Centre Hospitalier Universtaire of Montpellier for Tuberous Sclerosis
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Phenotype | 1 day
  Phenotype : Dermatological signs observed

SECONDARY OUTCOMES:
Genotype | 1day
  Genotype : TSC1, TSC2, mosaicism

CONTACTS AND LOCATIONS:
Overall Officials: Didier BESSIS, PhD, Principal Investigator — University Hospitals of Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC